CLINICAL TRIAL: NCT04774055
Title: A Combined Microdialysis and FDG-PET Study for Detection of Brain Injury in Comatose Survivors Resuscitated From Out-of-hospital Cardiac Arrest - a Pilot Study
Brief Title: A Combined Microdialysis and FDG-PET Study for Detection of Brain Injury After Cardiac Arrest
Acronym: COMA-PROTECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Simon Mölström, Consultant physician, Odense University Hospital
Other Study IDs: S-20150173 HLO
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Arrest; Brain Injuries
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain injury remains the leading cause of death in comatose patients resuscitated from OHCA. One of the most challenging aspects in the treatment of a post-cardiac arrest patient is the assessment of the extent of brain damage. Reliable, clinical measures of ongoing brain injury have potential to guide individualized treatment and potentially improve outcomes. Persistent candidate measures to fill this role is combined cerebral metabolism monitoring assessed by jugular bulb microdialysis (JBM) and positron emission tomography (PET) of 18-Fluor deoxyglucose ([F-18]-FDG). This multimodal neuromonitoring is cutting-edge technology used in a clinical setting

DETAILED DESCRIPTION:
Background Survival rates around 50 % are reported in comatose patients treated with hypothermia in Intensive Care Unit (ICU) after out-of-hospital cardiac arrest (OHCA). The high risk of ICU death is generally due to the primary hypoxic-ischemic insult, and subsequently secondary brain damage caused by prolonged insufficient cerebral blood flow (CBF), disturbed autoregulation, ischemia-reperfusion injury and compromised cerebral energy metabolism injury. Conclusive evidence of secondary cerebral ischemia following cardiac arrest has been elusive. Secondary injury is a significant determinant of neurologic outcome, and alleviating its deleterious effects is a mainstay of post-cardiac arrest management. This far, the clinicians still need more accurate monitoring methods to identify and manage potential reversible ongoing brain ischemia, and predicting early neurological outcome in the ICU. Methods measuring global brain ischemia and reflecting metabolic perturbations after resuscitation are needed for a more individualized post-resuscitation care-and target-driven therapy to improve patient outcome.

Jugular bulb microdialysis (JBM) allows global cerebral metabolic variables of the draining venous blood to be monitored continuously and provides data on substrate supply and metabolism at the cellular level in the brain. The ability to measure global brain metabolites concentration of glucose, pyruvate, lactate, lactate to pyruvate ratio (LPR), glutamate and glycerol at the bedside has provided the option of utilizing JBM as a clinical brain-monitor. High LPR > 30 is considered a robust indicator of anaerobic metabolism (low pyruvate) and is an independent predictor of mortality and unfavorable outcome in traumatic brain injury among patients monitored with MD (1-6).

Our group has recently published that I) metabolic monitoring in the jugular bulb is representative of the overall cerebral metabolism and can be used in the diagnosis of compromised global cerebral metabolism during cardiac surgery (7) and II) global JBM indicating isolated early brain injury was found after OHCA and consecutive resuscitation (study in press) III) preliminary JBM data indicates that approximately 30 % of comatose OHCA survivors (cerebral performance category 3-5, poor neurological outcome) are suffering from early secondary brain ischemia (8).

Further advances in the knowledge of cerebral metabolism have been achieved by applying positron emission tomography (PET) of 18-Fluor deoxyglucose ([F-18]-FDG) to OHCA patients, enabling cerebral metabolic rate of glucose CMRglc to be quantified (9-10). PET provides a global metabolic map of the whole brain but only for the duration of the scan. FDG-PET measurement is primarily a marker of glucose uptake, which cannot be used to determine the fate of this brain fuel. At the same time, the JBM variables have the potential of displaying several options regarding the fate of glucose and signs of metabolic crisis. It is in this context that the present study attempts to determine if there is a metabolic crisis due to ischemia or due to mechanisms other than ischemia by examining global brain tissue with combined positron emission tomography and jugular bulb microdialysis. The sensitivity of JBM to detect relevant secondary brain injury in cardiac arrest patients is further investigated through comparative imaging with PET-CT.

Aim The study aim to use 18-Fluorodeoxyglucose positron emission tomography (PET) combined with jugular bulb microdialysis to investigate pathophysiological brain derangements following cardiac arrest.

Endpoints Primary endpoint: The difference in overall CMRglc at day 0 and 3 after OHCA between neurological outcome groups

Secondary endpoints:

1. Correlation between JBM variables and the overall CMRglc on day 0 and 3 after OHCA.
2. Do the patterns of PET-verified global glucose metabolism reflect the early global neuro-metabolic pattern (ischemia/mitochondrial dysfunction) obtained by jugular bulb microdialysis following OHCA.

Method A prospective feasibility study designed to investigate pathophysiological brain derangements following cardiac arrest using combined 18-FDG-PET with jugular bulb microdialysis (JBM). Ten unconscious patients admitted to the ICU, with sustained return of spontaneous circulation after out-of-hospital cardiac arrest will be included. Assent will be obtained from the next of kin.

For detection of early global brain ischemia in the post-resuscitation phase jugular bulb microdialysis catheters will be implanted as fast as possible after ICU admission. Patients will be monitored for 96 hours or until arousal or withdrawal of life-sustaining therapy. Intravenous microdialysis catheters (CMA 67 IV 130 mm, membrane length 10 mm, MDialysis AB, Stockholm, Sweden) with 20 kDa molecular weight cut-off membranes enable the measurement of energy-related metabolites: glucose, lactate, pyruvate, LPR, glutamate and glycerol. The samples will be collected in microvials for analysis every one hour by enzymatic photometric techniques, and presented bedside.

FDG-PET will be obtained on day 0 and 3 after OHCA regardless of neurological status. Neurological outcome is assessed at hospital discharge according to the Cerebral Performance Category (CPC) scale: CPC 1 - no neurological deficit; CPC 2 - mild to moderate dysfunction; CPC 3 - severe dysfunction; CPC 4 - coma; and CPC 5 - death. CPC scores of 1 and 2 are considered as 'good' outcomes and a CPC 3-5 'poor' outcomes.

Limitations Lateralization in cerebral venous drainage may affect jugular bulb sampling. Although, the investigators use bedside ultrasound to identify the dominant jugular vein, and the JBM technique is applied to a condition producing strictly global cerebral injury and hypoxic ischemia. Clinicians are not blinded to data obtained bedside from jugular bulb microdialysis, so all outcome assessors will be blinded to minimize the risk of bias. Simultaneously cerebral blood flow cannot be estimated due to logistics and operational costs.

Expected clinical impact The mortality of patients who are admitted in a comatose state following successful resuscitation after cardiac arrest remains high. Combined JBM and FDG-PET have the clinical potential to provide novel insights in dynamic pathogenic metabolic patterns related to secondary brain injury. Combining these two technologies would, therefore, appear to be attractive aiming at exploring whether brain tissue after a period of global transient ischemia displays biochemical signs of ongoing ischemia. In the future, this multimodal approach might optimize brain metabolism and individualize the treatment of post-cardiac arrest patients suffering from secondary ischemia and potentially improve outcomes.

Project feasibility The research group has shown that metabolic monitoring in the jugular bulb is representative of the overall cerebral metabolism and can be used in the diagnosis of compromised global cerebral metabolism in a clinical setting. The next step is to combine jugular bulb microdialysis with FDG-PET in a pilot study to prove the feasibility of this novel combined technique.

Ethical justification

Participation in the study will not interfere with or delay routine diagnostic or therapeutic procedures. The ethical justification for participating in the COMA-PROTECT study is:

Knowledge of cerebral metabolism in comatose patients resuscitated after OHCA cannot be gained outside the acute setting.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA) of presumed cardiac cause
* Sustained return of spontaneous circulation (ROSC), defined as ROSC when chest compressions have not been required for 20 consecutive minutes and signs of circulation persist
* Unconsciousness (Glasgow Coma Scale (GCS) score of less than 8) after sustained ROSC
* Target temperature management (TTM) is indicated.

Exclusion Criteria:

* Conscious patient (GCS score of at least 8)
* Female of child-bearing potential, unless a negative human chorionic gonadotropin (hCG) test can rule out pregnancy within the inclusion window
* In-hospital cardiac arrest (IHCA)
* OHCA of presumed non-cardiac cause, such as after trauma, dissection/rupture of major artery or arrest caused by hypoxia (i.e., drowning, hanging, etc.)
* Known bleeding diathesis (medically induced coagulopathy does not exclude patient)
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute ischemic stroke
* Unwitnessed asystole
* Known limitations in therapy and do-not-resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose patients after OHCA admitted to the hospital with sustained return of spontaneous circulation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall CMRglc | Day 0 after cardiac arrest
  Cerebral metabolic rate of glucose (CMRglc)
Overall CMRglc | Day 3 after cardiac arrest
  Cerebral metabolic rate of glucose (CMRglc)

SECONDARY OUTCOMES:
Jugular bulb microdialysis (JBM) LP ratio | Day 0 after cardiac arrest
  Correlation between time-averaged (24 h) JBM lactate/pyruvate (LP) ratio and the overall CMRglc
JBM LP ratio | Day 3 after cardiac arrest
  Correlation between time-averaged (24 h) JBM LP ratio and the overall CMRglc

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mølstrøm, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Undecided